CLINICAL TRIAL: NCT04922879
Title: Early Lung Rehabilitation Care for Patients After Double Lung Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020--499
Record Dates: First submitted 2021-06-01; First posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Pulmonary Disease
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Intervention Model Description: experience summary
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individualized lung rehabilitation programme (Experimental): Early respiratory function training, reasonable oxygen therapy to prevent hypoxemia, Positive pressure vibration training to promote coughing ability recovery, early exercise, Health education and psychological support.
  Interventions: Behavioral: Individualized lung rehabilitation

INTERVENTIONS:
Behavioral: Individualized lung rehabilitation — Early respiratory function training, reasonable oxygen therapy to prevent hypoxemia, Positive pressure vibration training to promote coughing ability recovery, early exercise, Health education and psychological support.

SUMMARY:
Develop appropriate individual programs for patients to implement lung rehabilitation safely and effectively.

DETAILED DESCRIPTION:
Early respiratory function training, reasonable oxygen therapy to prevent hypoxemia, Positive pressure vibration training to promote coughing ability recovery, early exercise, Health education and psychological support.

ELIGIBILITY:
Inclusion Criteria:

* Patients after double lung transplantation; informed consent

Exclusion Criteria:

* unstable condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
ICU hospital stay | 1 year
  the stay time spent in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Fei Zeng, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- SAHZhejiangU, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No